CLINICAL TRIAL: NCT03166696
Title: The Registry and Follow-up of Patients With Acute Myocardial Infarction or Acute Cerebral Infarction
Brief Title: Acute Myocardial Infarction and Acute Cerebral Infarction (AMIAC) Registry and Follow-up
Acronym: AMIAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Shi, Professor, Guangdong Provincial People's Hospital
Other Study IDs: 20170309
Record Dates: First submitted 2017-05-18; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Myocardial Infarction; Cerebral Infarction; Chronic Kidney Diseases; Mortality
MeSH Terms: conditions — Myocardial Infarction; Cerebral Infarction; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute cerebral infarction: the registry and follow up of consecutive patients who were admitted and diagnosed with acute cerebral infarction
- acute myocardial infarction: the registry and follow up of consecutive patients who were admitted and diagnosed with acute myocardial infarction

SUMMARY:
A registry of consecutive patients who were admitted and diagnosed with acute myocardial infarction or acute cerebral infarction were conducted at the Guangdong General Hospital or the First Affiliated Hospital of Guangzhou University of Chinese Medicine, Yue Bei People's Hospital, China, between January 2000 and December 2016. The adverse clinical outcomes, including all-cause mortality, were followed from the date of admission for acute myocardial infarction or acute cerebral infarction until study end (December 31, 2016). All-cause mortality, including the date of death, was identified from the electronic hospitalization data, phone follow-up, and confirmed by the household registration (HUKOU) system, a record of registration required by law in China. Baseline characteristics, including major treatment of acute myocardial infarction or acute cerebral infarction, estimated glomerular filtration rate (eGFR) and proteinuria, were collected. Demographic data were determined from the electronic hospitalization data and electronic hospital discharge records. All comorbid conditions were identified using International Statistical Classification of Diseases, Tenth Revision (ICD-10), coding algorithms applied to electronic physician claims and electronic hospital discharge records. Life style (smoking), treatment regimen at discharge, including angiotensin-converting enzyme inhibitor (ACEI), angiotensin II receptor blocker (ARB), were determined from the electronic hospitalization data.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients who were admitted and diagnosed with acute myocardial infarction or acute cerebral infarction

Exclusion Criteria:

* lacunar infarction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the consecutive patients who were admitted and diagnosed with acute myocardial infarction or acute cerebral infarction at the Guangdong General Hospital or the First Affiliated Hospital of Guangzhou University of Chinese Medicine, Yue Bei People's Hospital, China, between January 2000 and December 2016.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2000-01-03 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | follow up until the study end (May 2018,Anticipated)
  all-cause mortality

SECONDARY OUTCOMES:
kidney outcome | follow up until the study end (May 2018,Anticipated)
  ESRD or 50%eGFR decline

CONTACTS AND LOCATIONS:
Overall Officials: Liming Yao, M.D., Study Director — Guangdong Provincial People's Hospital
Locations (3):
- China (3):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - the First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong

IPD SHARING:
Plan to Share IPD: No